CLINICAL TRIAL: NCT00121758
Title: Randomised Double Blinded Phase II AIDS Vaccine Study Comparing Immunogenicity and Safety of 3 Doses of Lipopeptide (LIPO-5) Versus Placebo in Non Infected HIV Volunteers (ANRS VAC 18)
Brief Title: AIDS Vaccine Study Comparing Immunogenicity and Safety of 3 Doses of Lipopeptides Versus Placebo in Non Infected HIV Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004-000233-10; ANRS VAC18
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: HIV Vaccines; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: LIPO-5

SUMMARY:
This study will test the safety and immune response to an experimental HIV vaccine, LIPO-5, in healthy volunteers. LIPO-5 contains 5 lipopeptides from gag, nef and pol corresponding to more than 50 epitopes. LIPO-5 has been shown to be immunogenic and well tolerated in a first phase I trial in non-HIV infected volunteers. Lower doses of each peptide could have a similar immunogenicity.

DETAILED DESCRIPTION:
The aims of HIV lipopeptide vaccination approach are to improve cell mediated immune responses in order to obtain strong, long lasting and polyepitopic responses and to focus these responses on highly conserved and immunogenic epitopes.

Lipopeptides are chemically synthetized peptides, bearing HIV epitopes, covalently bound to a fatty acid moiety, a monopalmtoyl chain in this case. This lipid chain produces internalization of the lipopeptide into the cytoplasm of the antigen presenting cells. Combinations of several lipopeptides containing sequences from different HIV proteins are used in vaccination trials in order to increase polyepitopic responses. Lipopeptides have been synthetized by the French National Agency for Research on AIDS and Viral Hepatitis (ANRS) preventive program by the group of Helen Gras following a long and meticulous work of epitope screening performed by the team of Jean-Gérard Guillet at the Cochin Institute in Paris. The epitopes were selected on the basis of their strong affinity for HLA class I molecule, on their ability to form a stable complex with these molecules, and on the capacity of these epitopes to be recognized by T cells. The selected peptides are those containing the richest array of epitopes and those most frequently recognized by HIV infected patients. Each peptide has a length of 23 to 32 amino acids (AA).

Different types of lipopeptides constructs have been tested in humans. Among these constructs, LIPO-5 contains 5 lipopeptides from gag, nef and pol corresponding to more than 50 epitopes. LIPO-5 has been shown to be immunogenic and well tolerated in a first phase I trial in non-HIV infected volunteers. Lower doses of each peptide could have a similar immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers selected by ANRS (French National Agency for Research on AIDS and Viral Hepatitis)
* For woman of child-bearing age: use of effective contraception
* Ability to sign informed consent
* Beneficiary subjects of social security regimen-- Hepatitis B, hepatitis C, HIV, HTLV1 infection and syphilis negative
* Hemoglobin over 12.5 g/dl for women and over 13.5 g/dl for men

Exclusion Criteria:

* Previous participation in an HIV clinical trial
* Volunteers with risk to contract HIV infection during the trial
* Previous vaccination in the last month, and volunteers requiring vaccination during the trial
* Gift of blood in the last 2 months
* Eczema, urticaria
* Medical history of food allergy, Lyell or Stevens Johnson syndrome and aggravated asthma
* Previous (last 6 months) or ongoing administration of immunological treatment, chemotherapy, radiotherapy or corticosteroid
* Medical history of autoimmune disease
* Clinical or biological aftermath of previous disease
* Medical history of uveitis
* Transfusion in the last 6 months

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with CD8 immune response on ELISPOT IFN-gamma at week (W) 48

SECONDARY OUTCOMES:
Local and general adverse events
Percentage of subjects with CD4 immune response against different peptides of LIPO-5
Percentage of subjects with sustained response at week 48
Percentage of subjects with response against more than 1 peptide (multiepitopic response)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Salmon, MD, Principal Investigator — Hopital Cochin Paris. Centre des essais vaccinaux Cochin Pasteur; Christine Durier, Study Chair — Inserm SC10
Locations (1):
- CIC de Vaccinologie Cochin Pasteur, Paris, France

REFERENCES:
- [Derived] Richert L, Hue S, Hocini H, Raimbault M, Lacabaratz C, Surenaud M, Wiedemann A, Tisserand P, Durier C, Salmon D, Lelievre JD, Chene G, Thiebaut R, Levy Y; ANRS Vaccine Network/Vaccine Research Institute. Cytokine and gene transcription profiles of immune responses elicited by HIV lipopeptide vaccine in HIV-negative volunteers. AIDS. 2013 Jun 1;27(9):1421-31. doi: 10.1097/QAD.0b013e32835f5b60. PMID 23759749
- [Derived] Salmon-Ceron D, Durier C, Desaint C, Cuzin L, Surenaud M, Hamouda NB, Lelievre JD, Bonnet B, Pialoux G, Poizot-Martin I, Aboulker JP, Levy Y, Launay O; ANRS VAC18 trial group. Immunogenicity and safety of an HIV-1 lipopeptide vaccine in healthy adults: a phase 2 placebo-controlled ANRS trial. AIDS. 2010 Sep 10;24(14):2211-23. doi: 10.1097/QAD.0b013e32833ce566. PMID 20625264